Comparing EEG patterns in different age groups during general anesthesia with sevoflurane.

NTC number: NCT03559504

Date: 28/7/2018

## **STATISTICAL PLAN:**

Statistical analyses will be performed with a statistical package (SPSS version 21.0; SPSS, Chicago, IL) and Microsoft excel. All data will be presented as mean  $\pm$  sd. Demographic data will be compared by using standard t-tests; comparison of incidence data between groups performed by using Fisher's exact tests. A P value < 0.05 will be considered significant.

Data related to non-invasive blood pressure, heart rate, respiration rate, oxygen saturation, EEG waves frequencies, end tidal volume of sevoflurane and BIS values will be recorded. These data will be analyzed every 1min for the first 10mins during maintenance of anesthesia with 1.0 MAC sevoflurane. Data collection will be first recorded after tracheal intubation. The raw EEG wave will be recorded by means of a Universal Serial Bus (USB) which will later be analyzed and processed offline.

EEG waves, BIS values and Et sevoflurane will be collected every 1minute for a period of 10 minutes at T1,T2,T3,T4,T5,T6,T7,T8,T9,T10.

Non-invasive blood pressure, heart rate, respiration rate and oxygen saturation values will be recorded every 3 minutes for the same period (10minutes).